CLINICAL TRIAL: NCT00962442
Title: N-Acetylcysteine for the Treatment of Alcoholic Hepatitis: a Belgian Multicenter Randomised Trial
Brief Title: N-Acetylcysteine in Severe Acute Alcoholic Hepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Olivier Le Moine, MD, PhD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAH-LYSO
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis; N-Acetylcysteine; enteral nutrition; oxidative stress; severe acute alcoholic hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nutritional support + N-Acétylcysteine (Active Comparator): N-Acétylcysteine 300 mg/kg intravenously for 14 days Beside usual meals, patients must receive at least 27 kcal/kg/day enteral nutrition for 14 days
  Interventions: Drug: N-Acetylcysteine
- nutritional support + placebo (Placebo Comparator): placebo perfusion for 14 days Beside usual meals patients must receive at least 27 kcal/kg/day enteral nutrition for 14 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 300 mg/kg for 14 days, intravenously
  Arms: nutritional support + N-Acétylcysteine
Drug: placebo — Glucosé 5% perfusion for 14 days, intravenously
  Arms: nutritional support + placebo

SUMMARY:
Acute alcoholic hepatitis (AAH) is the most severe form of alcoholic liver disease (ALD) and is associated with a high risk of dying in the short term. Corticosteroids are generally recommended in patients with severe AAH, but its use is still controverted and contraindicated in case of active infection or gastrointestinal bleeding. Therefore, alternative therapeutic options are needed.Ethanol consumption results in the depletion of endogenous antioxidant capabilities and patients with ALD have evidence of antioxidant deficiencies.Due to its effects on glutathion stores restoration and as such the limitation of the oxidative stress and its good tolerance and safety profile, N-acetylcysteine (NAC) is an attractive agent for the treatment of AAH.In this context, we hypothesized that NAC might be beneficial in severe AAH.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven alcoholic hepatitis
* Severe disease defined by a Maddrey score superior to 32

Exclusion Criteria:

* Neoplastic disease compromising 6 months survival
* HIV patients
* Hepatorenal syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-09; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Six months survival

SECONDARY OUTCOMES:
Rate of infections, clinical and biological parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium